CLINICAL TRIAL: NCT04658004
Title: Clinical Trial for the Safety and Efficacy of NKG2D CAR-T Cell Therapy for Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Brief Title: NKG2D CAR-T Cell Therapy for Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKG2D-001
Record Dates: First submitted 2020-10-22; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; CAR T-cell therapy; NKG2D
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of NKG2D CAR T-cells (Experimental)
  Interventions: Drug: NKG2D CAR T-cells

INTERVENTIONS:
Drug: NKG2D CAR T-cells — Each subject receive NKG2D CAR T-cells by intravenous infusion
  Other Names: NKG2D CAR-T cells injection

SUMMARY:
A Study of NKG2D CAR-T Cell Therapy for Patients With Relapsed and/or Refractory Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory NKG2D ligand positive acute myeloid leukemia. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 36 patients will be enrolled. Primary objective is to explore the safety,main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of NKG2D ligand positive AML per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Myeloid Leukemia (2016.v1);
2. Relapsed or refractory NKG2D ligand positive AML (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is less than 12 months;
   3. Ineffectively after first or multiple remedial treatments;
   4. 2 or more relapses;
3. The number of primordial cells in bone marrow is > 5% (by morphology), and/or > 0.01% (by flow cyto metry);
4. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
5. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
6. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
7. Estimated survival time ≥ 3 months;
8. ECOG performance status 0 to 2;
9. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance,epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
7. Previously treated with any CAR-T cell product or other genetically modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after NKG2D targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after NKG2D targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Acute Myeloid Leukemia (AML), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 1, 3, 6, 12, 18 and 24
AML, Overall survival (OS) | Up to 2 years after NKG2D CAR-T cells infusion
  . AML, Overall survival (OS) From the first infusion of NKG2D CAR-T cells to death or the last visit
AML, Event-free survival (EFS) | Up to 2 years after NKG2D CAR-T cells infusion
  From the first infusion of NKG2D CAR-T cells to the occurrence of any event, including death, relapse or gene relapse disease progression (any one occurs first), and the last visit
Quality of life | :At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No